CLINICAL TRIAL: NCT04781972
Title: Multimodal Brain Imaging of the Neural Effects of Methylphenidate in Patients With ADHD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00276357
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: ADHD - Combined Type
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: This is a double-blind cross over of a single dose of methylphenidate (10mg or 15mg) and matching placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylphenidate first (Experimental): Single oral dose of methylphenidate (10mg or 15 mg) and then matching placebo after washout period of one week.
  Interventions: Drug: Methylphenidate; Drug: Placebo
- Placebo first (Placebo Comparator): Matching placebo and then single oral dose of methylphenidate (10mg or 15 mg) after washout period of one week.
  Interventions: Drug: Methylphenidate; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — single dose of 10 mg or 15 mg
Drug: Placebo — Matching placebo

SUMMARY:
The investigators' goal is to develop neuroimaging biomarkers to predict response to treatment with methylphenidate, which then can be used in the development of novel pharmacological treatments for attention-deficit/hyperactivity disorder (ADHD). The overall objective of this study is to measure the changes in task-related neural activity related to symptoms of ADHD (measured by functional MRI) and brain glutamate levels (measured by magnetic resonance spectroscopy, MRS) after treatment with methylphenidate (MPH). This will be a double-blind crossover of methylphenidate and placebo in adults with ADHD. Participants will complete neuropsychological testing along with fMRI and MRS scans after a single dose of each treatment.

ELIGIBILITY:
Inclusion Criteria:

* right handed

Exclusion Criteria:

* pregnant or breast feeding
* past or current neurological disorder
* non-ADHD cause of cognitive impairment
* uncontrolled medical disorder
* head trauma with loss of consciousness in the last year or any evidence of functional impairment due to and persisting after head trauma
* having an adverse reaction to methylphenidate, or other stimulant medication
* having a contraindication to MRI
* current smoking

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
BOLD signal during response inhibition | Approximately 90 minutes after dose
  BOLD signal (brain activity during fMRI, arbitrary units) in the anterior cingulate cortex during response inhibition.
Glutamate level in the anterior cingulate cortex | Approximately 2 hours after dose
  Glutamate level (measured by MRS, institutional units) in the anterior cingulate cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Bigos, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No